CLINICAL TRIAL: NCT03703154
Title: Alterations in Cognitive Function and Cerebral Blood Flow After Conversion From Immediate Release Tacrolimus to Slow Release Envarsus
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Aditi Gupta, MD, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY00142282
Record Dates: First submitted 2018-09-13; First posted 2018-10-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 6 teaspoons of blood will be collected at each of the two visits and stored for future research (optional). This blood will be stored in the University of Kansas Kidney Institute Freezer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Arm: The patients in the study arm will be converted from immediate release Tacrolimus to Envarsus. After obtaining informed consent, participants will undergo baseline tests for cognitive function and cerebral blood flow. After 12 weeks, cognition and brain blood flow will be assesses again in all enrolled patients.
  Interventions: Drug: Envarsus
- Control Arm: Patients in the control arm will remain on the immediate release Tacrolimus. After obtaining informed consent, participants will undergo baseline tests for cognitive function and cerebral blood flow. After 12 weeks, cognition and brain blood flow will be assesses again in all enrolled patients.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Envarsus — Patients will then be randomized in the ratio of 2:1 with 20 being in the study arm and 10 in the control arm. Envarsus will be prescribed by the transplant team per conversion guidelines. The transplant team will monitor drug levels, per the dosing guidelines.
  Groups: Study Arm
Drug: Tacrolimus — The patient's physician will prescribe drug according to standard practice.
  Other Names: Prograf
  Groups: Control Arm

SUMMARY:
The purpose of this study is to learn if conversion from immediate release tacrolimus to Envarsus improves cerebral blood flow, brain blood flow response to exercise, and cognition.

DETAILED DESCRIPTION:
Each patient will have two study assessments: one at baseline and another one at 12 weeks after the baseline assessment. Each assessment may be divided into 2 visits to accommodate the MRI and TCD (Transcranial Doppler ultrasound). Detailed medical history will be extracted from the patients' medical records, interviews and questionnaires. We will obtain brain MRI (without gadolinium contrast) in enrolled patients. Neuropsychological test (NP) tests will include a standard battery to detect subclinical changes in cognition which can be missed by screening tests like the mini mental state exam.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 85 years
* English speaking (NP tests will be in English);
* able to sign informed consent
* able to arrange transportation to and from study sites
* without acute stroke, concussion or traumatic brain injury
* received a kidney transplant at least 12 weeks before recruitment
* stable kidney function with serum creatinine <3mg/dl

Exclusion Criteria:

* are claustrophobic or have other contra-indication for MRI
* have hearing or visual impairment
* are unable to read, write, speak or understand English
* have uncontrolled psychosis or seizure disorder or are currently using antipsychotics or anti-epileptics
* dual organ transplant
* oxygen-dependent chronic obstructive pulmonary disease
* diagnosis of dementia
* unable to perform exercise on the Nustep (muscle weakness or cardiac safety concern)
* uncontrolled blood pressure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the KUMC kidney transplant clinic. Both male and female kidney transplant recipients aged 18 to 85 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function using a battery of neuropsychological tests | Change from Baseline to Week 12
  Battery aggregate scores include such tests as: Mini Mental Sate Exam, Montreal Cognitive Assessment, Digit Span, Logical Memory, Category Fluency, Trail Making, Digit Symbol, Block Design, Stroop, Buschke Free and Cued Reminding Test.
Change in cerebral blood flow | Change from Baseline to Week 12
  including brain blood flow response curve to exercise or cerebral reactivity

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Gupta, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States